CLINICAL TRIAL: NCT05044130
Title: Postprandial Hepatic Fatty Acid Metabolism During Oral High-fat Mixed-meal Challenge Test in Patients With Type 2 Diabetes With and Without NAFLD
Brief Title: Postprandial VLDL-triglyceride Metabolism in Type 2 Diabetes Patients With and Without NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Diabetes Academy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 01072021
Record Dates: First submitted 2021-09-04; First posted 2021-09-14 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: NAFLD; Type 2 Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 Diabetes with NAFLD (Active Comparator): Patients with Type 2 Diabetes with NAFLD
  MR spectroscopy verified steatosis
  Interventions: Dietary Supplement: High-fat mixed-meal tolerance test (HF-MMTT)
- Type 2 Diabetes without NAFLD (Active Comparator): Patients with Type 2 Diabetes without NAFLD
  MR spectroscopy verified no steatosis
  Interventions: Dietary Supplement: High-fat mixed-meal tolerance test (HF-MMTT)

INTERVENTIONS:
Dietary Supplement: High-fat mixed-meal tolerance test (HF-MMTT) — The test meal consists of a standardized HF-MMTT (791 cal) with 197 g cream (38 % fat), 18 g sugar and 1 g vanilla sugar for taste (75 g fat, 25 g carbohydrate and 4 g protein)

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) covers a spectrum from simple reversible hepatic steatosis to inflammation and fibrosis termed steatohepatitis (NASH). The mechanisms behind why some subjects progress from NAFLD to NASH are not clear and the responsible mechanism for storage of excess amounts of liver fat in patients with NAFLD are poorly understood.

Patients with type 2 diabetes mellitus (T2D) and abdominally obese subjects very often have accumulation of liver fat (NAFLD).

T2D is also associated with abnormal lipid metabolism (dyslipidemia), including free fatty acids (FFA), hypertriglyceridemia and excessive postprandial hyperlipidemia which increases the risk of ischemic cardiovascular disease (CVD) and heart failure.

In healthy, insulin sensitive subjects the postprandial increase in triglycerides (TG) is primarily caused by meal derived chylomicrons, whereas endogenously produced TG (VLDL-TG) and decreased peripheral TG clearance only becomes quantitatively important in insulin resistant subjects .Thus, postprandial lipidemia in T2D results from both chylomicronemia as well as a reduction in both insulin mediated suppression of VLDL-TG secretion and lipoprotein lipase (LPL) mediated peripheral clearance. A recent study demonstrated that the ability of insulin to suppress hepatic VLDL-TG after a fat-enriched meal and the duration of the postprandial hyperlipidemia was similar in patients with T2D compared with age- and BMI matched individuals without T2D, indicating that the degree of insulin mediated VLDL-TG secretion and hyperlipidemia primarily depends on insulin sensitivity and not the presence of T2D diabetes per se.

In these studies, the investigators want to examine the effect of a fat enriched mixed-meal on hepatic VLDL-TG handling and adipose storage capacity in patients with T2D with and without NAFLD. Investigators will address these questions using carboxyl-14C triolein labeled VLDL-TG, magnetic resonance (MR) spectroscopy of liver, muscle and fat biopsies in combination with state-of-the art muscle and adipose tissue enzyme kinetics, gene- and protein expression.

The overarching goals are to define abnormalities and differences between patients with T2D with and without NAFLD in terms of hepatic lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 Diabetes with and without NAFLD (steatosis FF% > 5,6% on MR spectroscopy for NAFLD and NASH groups)

Exclusion Criteria:

* Active smoking
* Comorbidity other than hypertension and hyperlipidemia
* Fixed medical drug consumption (including insulin) except statins and anti-diabetic medications. However, statins must be paused 2 weeks before the examination date and other antidiabetic medication on examination date.
* Patients with cancer or former cancer patients
* Blood donation within the last 3 months prior to the study
* Participation in experiments involving radioactive isotopes within the last 3 months
* Alcohol abuse (over 21 items per week for men and over 14 for women)
* Pregnancy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
VLDL-triglyceride secretion - Ex vivo labeled VLDL - [14C]-triolein tracer technique. | 1 day
  (μmol/min)
VLDL-triglyceride uptake in muscle - Measurement of fatty acid concentration and specific activity in muscle biopsies | 1 day
  (percent)
VLDL-triglyceride uptake in adipose tissue - Measurement of fatty acid concentration and specific activity in adipose tissue biopsies | 1 day
  (percent)

SECONDARY OUTCOMES:
VLDL-triglyceride oxidation - Oxidation is measured by specific activity in exhaled air. | 1 day
  (μmol/min)
Adipose cell size measurement | 1 day
  (μl)
Insulin sensitivity | 1 day
  (mg/kg/min)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus N, Denmark